CLINICAL TRIAL: NCT04393727
Title: Transfusion of Convalescent Plasma for the Early Treatment of pneumonIa Due to SARSCoV2: a Multicenter Open Label Randomized Control Trial
Brief Title: Transfusion of Convalescent Plasma for the Early Treatment of Patients With COVID-19
Acronym: TSUNAMI
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was stopped because the Promoter was changed and a new study on convalescent plasma promoted by AIFA was started in Italy.
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Francesco Menichetti, Professor, Azienda Ospedaliero, Universitaria Pisana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TSUNAMI
Record Dates: First submitted 2020-05-16; First posted 2020-05-19 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: COVID; SARS-CoV 2
Keywords: covid-19; SARS-CoV2; pneumonia; convalescent plasma
MeSH Terms: conditions — COVID-19; Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients in the intervention group will receive 200 cc of convalescent plasma
  Interventions: Biological: CONVALESCENT PLASMA
- Control (No Intervention): Patients will continue to receive standard therapy

INTERVENTIONS:
Biological: CONVALESCENT PLASMA — Convalescent plasma will be collected by healthy donors, cured by COVID-19 and, after standard preparation and dosage of neutralizing antibodies, will be administered to patients with SARS-CoV2 pneumonia
  Arms: Intervention

SUMMARY:
No specific therapeutic agents or vaccines for COVID-19 are available. Several therapies, are under investigation, but the antiviral efficacy of these drugs is not yet known. The use of convalescent plasma was recommended as an empirical treatment during outbreaks of Ebola virus in 2014, and a protocol for treatment of Middle East respiratory syndrome coronavirus with convalescent plasma was established in 2015. Accordingly, we hypothesized that use of convalescent plasma transfusion could be beneficial in patients infected with SARS-CoV-2.

This is a multicenter prospective randomized clinical trial to evaluate safety and efficacy of early use of convalescent plasma in patients with SARS-CoV2 pneumonia.

Primary endpoint will be the efficacy, evaluated as the need of invasive mechanical ventilation defined by PaO2/FiO2 ratio <150.

Secondary endpoints will be: mortality rates, time to invasive mechanical ventilation, time to virological cure, length of hospital stay, toxicity.

Patients with SARS-CoV2 pneumonia not requiring mechanical ventilation (both non invasive and invasive) will be randomized 1:1 to receive or not convalescent plasma. Patients in the plasma group will receive 200 ml of convalescent plasma, continuing already administered standard therapy, while patients in the control group will continue to receive the standard therapy. A rescue therapy will be allowed in case of clinical worsening.

Patients will be followed-up until 30 days from randomization.

DETAILED DESCRIPTION:
This is a multicenter prospective randomized open-label clinical trials. Patients with pneumonia due to SARS-CoV-2 will be included and randomized to receive or not convalescent plasma.

Convalescent plasma will be collected by cured patients with previous diagnosis of COVID-19. More specifically, inclusion and exclusion criteria for donors will be the following.

Inclusion criteria for donors:

* age > 18 and <60 years
* confirmed diagnosis of COVID-19: PCR on nasopharynx swab or positive IgG
* presence of 2 negative nasopharynx swabs for patients with previous positive swab and presence of 1 negative nasopharynx swab for patients with positive IgG

Exclusion criteria for donors:

* age < 18 ys or >60 ys
* other conditions that controindicate blood donation

Collected plasma will undergo all procedures for blood preparation. Plasma will be tested with enzyme-linked immunosorbent assay (ELISA) and neutralizing antibody titers.

Patients eligible for the study will be selected among hospitalized patients with SARS-CoV2 pneumonia. More specifically, the following criteria will used for inclusion in the study.

Inclusion criteria for recipients:

* age >18 ys
* confirmed diagnosis of SARS-CoV2 pneumonia
* PaO2/FiO2 200-350

Exclusion criteria for recipients:

* PaO2/FiO2 <200
* need of non invasive or invasive mechanical ventilation

Patients will be randomized 1:1 to receive or not convalescent plasma. All patients will be followed-up for 30 days after randomization.

Primary endpoint will be the need of mechanical ventilation, defined as PaO2/FiO2 <150.

ELIGIBILITY:
Inclusion Criteria:

* Any gender
* Age > 18 years on day of signing informed consent
* Informed written consent for participation in the study
* Virological diagnosis of SARS-CoV-2 infection (real-time PCR)
* Hospitalized due to clinical instrumental diagnosis of pneumonia
* PaO2/FiO2 ratio 200-350

Exclusion Criteria:

* mechanical ventilation (both invasive and non-invasive)
* PaO2/FiO2<200
* known hypersensitivity to immunoglobulin or blood components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Need of invasive mechanical ventilation | 30 days
  Need of invasive mechanical ventilation defined as PaO2/FiO2 <150

SECONDARY OUTCOMES:
Mortality rates | 30 days
  Thirty-day mortality rates
Time to invasive mechanical ventilation | 30 days
  Days from randomization to invasive mechanical ventilation
Time to virologic cure | 30 days
  Days from randomization to virologic cure defined as 2 consecutive negative nasopharynx swabs
Length of hospital stay | 30 days
  Days from randomization to discharge or death
Adverse events | 30 days
  Occurrence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Menichetti, Principal Investigator — Azienda Ospedaliero, Universitaria Pisana
Locations (1):
- Azienda Ospedaliero Universitaria Pisana, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shen C, Wang Z, Zhao F, Yang Y, Li J, Yuan J, Wang F, Li D, Yang M, Xing L, Wei J, Xiao H, Yang Y, Qu J, Qing L, Chen L, Xu Z, Peng L, Li Y, Zheng H, Chen F, Huang K, Jiang Y, Liu D, Zhang Z, Liu Y, Liu L. Treatment of 5 Critically Ill Patients With COVID-19 With Convalescent Plasma. JAMA. 2020 Apr 28;323(16):1582-1589. doi: 10.1001/jama.2020.4783. PMID 32219428